CLINICAL TRIAL: NCT03083340
Title: Implementation of a Self-Help Depression Program Among Orthopedic Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility concerns regarding recruitment
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-08-0089
Record Dates: First submitted 2017-02-24; First posted 2017-03-20 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: MDD

STUDY DESIGN:
Intervention Model Description: Deprexis consists of 10 content modules representing different psychotherapeutic approaches, plus one introductory and one summary module, each of which can be completed in 10 to 60 minutes, depending on the user's reading speed, interest, motivation, and individual path through the program (Meyer, et al., 2009).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deprexis (Experimental): Participants will complete 8 weeks of online treatment via a web-based program, Deprexis.
  Interventions: Behavioral: Deprexis

INTERVENTIONS:
Behavioral: Deprexis — Participants will complete an 8 week self-help computerized treatments through a web-based online Deprexis program.

SUMMARY:
The proposed study addresses the potential utility of providing an accessible self-help intervention for patients in a medical setting with an estimated diagnosis of MDD. Specifically, the study will explore whether a) such an intervention can be effectively implemented in a primary care setting and b) patients originally seeking medical attention for an orthopedic problem will be willing to seek psychological treatment and, c) improvement in depression symptoms will lead to improvement in upper and lower extremity functioning.

DETAILED DESCRIPTION:
The present project will be an open-label trial to assess the feasibility and acceptability of a self-help intervention among a sample of orthopedic patients. In addition to monitoring the effectiveness of the Deprexis program on depressive symptoms, the proposed project will assess whether a reduction in depressive symptoms will be associated with improvement on patient reported orthopedic impairment. The investigators will enroll 50 adults and the participants will be given the opportunity to participate in 8 weeks of the web-based online Deprexis program.

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 18 years who present to a surgeon with an upper or lower extremity injury or disability at a participating center (see attached list)
* A level of clinical depression more than minimal symptoms as defined by a score ≥ 10 on the Patient Health Questionnaire-9 (PHQ-9)
* Willing and able to provide informed consent and comply with the protocol

Exclusion Criteria:

* Injury or illness best treated with prompt surgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Proof of Concept - Acceptability measured by number of eligible participants that choose to participate | 8 weeks
  The primary outcome will be the level of acceptability of the intervention as measured by the number of eligible participants who chose to participate in the intervention.
Proof of Concept - Acceptability measured by number of modules completed on the online program | 8 Weeks
  The primary outcome will be the level of acceptability of the intervention as measured by number of completed modules on the online Deprexis program.
Proof of Concept - Acceptability measured by qualitative feedback | 8 Weeks
  The primary outcome will be the level of acceptability of the intervention as measured by qualitative feedback following the intervention created by the investigators on how acceptable the study was for the participant.
Proof of Concept - Feasibility measured by number of eligible participants that choose to participate | 8 Weeks
  The primary outcome will be the level of feasibility of the intervention as measured by he number of eligible participants who chose to participate in the intervention.
Proof of Concept - Feasibility measured by number of modules completed on the online program | 8 Weeks
  The primary outcome will be the level of acceptability of the intervention as measured by number of completed modules on the online Deprexis program.
Proof of Concept - Feasibility measured by qualitative feedback | 8 Weeks
  The primary outcome will be the level of acceptability of the intervention as measured by qualitative feedback following the intervention created by the investigators on how acceptable the study was for the participant.

SECONDARY OUTCOMES:
Level of Improvement of Depression (by scores on the PHQ-9) | 8 weeks
  Secondary outcome measures will be the level of depressive symptoms as evidenced by scores on the PHQ-9.
Level of Improvement of Functioning (by scores on the PROMIS Physical Function CAT) | 8 weeks
  Secondary outcome measure will be the level of improvement in upper and lower extremity function as measured by scores on the PROMIS Physical Function CAT.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No